CLINICAL TRIAL: NCT05092061
Title: Acute and Chronic Effects of Two Different Types of Resistance Training on Cardiometabolic Health in Adults With Obesity
Brief Title: Resistance Training in Adults With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 246888
Record Dates: First submitted 2021-09-20; First posted 2021-10-25 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Overweight and Obesity
Keywords: Exercise therapy; Muscular strength; Resistance training; Fitness testing; Healthy lifestyle
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The study will consist of both a crossover study model (acute phase) and parallel model (chronic phase).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-repetition resistance training (Experimental): The participants will undergo a full-body resistance training protocol with moderate repetitions (6-12), moderate load (70-85% of 1RM), and moderate rest between sets (60-90s). Training will be undertaken three times per week.
  Interventions: Other: Moderate-repetition resistance training
- High-repetition resistance training (Experimental): The participants will undergo a full-body resistance training protocol with high repetitions (15+), low load (<60% of 1RM), and short rest between sets (30s). Training will be undertaken three times per week.
  Interventions: Other: High-repetition resistance training

INTERVENTIONS:
Other: Moderate-repetition resistance training — Will undertake resistance training with moderate loads, and moderate repetitions 3 times per week for 7 weeks.
  Arms: Moderate-repetition resistance training
Other: High-repetition resistance training — Will undertake resistance training with low loads, and high repetitions 3 times per week for 7 weeks.
  Arms: High-repetition resistance training

SUMMARY:
The purpose of this project is two-fold: (1) to assess if two different resistance training protocols elicit different responses in the acute phase and (2) to assess if the same two different protocols will elicit different long-term responses on muscular strength, body composition and cardiometabolic health. The project will include 30 adults with obesity (defined as BMI ≥ 30 or abdominal obesity according to the International Diabetes Federation). In the acute phase blood lactate, heart rate, enjoyment and perceived exertion will be assessed after the two resistance training protocols. In addition, the mean 24-h blood glucose concentration after exercise will be compared between the two protocols.

For the long-term effects blood markers of cardiometabolic health, blood pressure, body composition, objectively measured physical activity and physical fitness will be assessed before and after the intervention. Also, perceived health-related quality of life will be assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI ≥ 30) or
* Central obesity (defined according to the International Diabetes Federation).

Exclusion Criteria:

* Unstable angina
* recent cardiac infarction (last 4 weeks)
* uncompensated heart failure
* severe valvular illness
* pulmonary disease
* uncontrolled hypertension
* kidney failure
* orthopaedic/neurological limitations
* cardiomyopathy
* planned operations during the research period
* participation in a parallel study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | 7 weeks

SECONDARY OUTCOMES:
Fasting glucose | 7 weeks
Blood lipid concentration | 7 weeks
C-reactive protein | 7 weeks
Systolic blood pressure | 7 weeks
Diastolic blood pressure | 7 weeks
Body fat | 7 weeks
  Measured by bioelectrical impedance (InBody 770)
Fat-free mass | 7 weeks
  Measured by bioelectrical impedance (InBody 770)
Body mass | 7 weeks
  Measured by bioelectrical impedance (InBody 770)
Visceral fat area | 7 weeks
  Measured by bioelectrical impedance (InBody 770)
Waist circumference | 7 weeks
VO2max (maximal aerobic capacity) | 7 weeks
Rate of force development | 7 weeks
  Measured by Kistler force plate
Muscular strength (1RM) | 7 weeks
  Leg press and bench press
Muscular endurance | 7 weeks
  Maximum number of repetitions using 50% of 1-RM
Physical activity | Baseline (before intervention), 4 and 7 weeks.
  Assessed at three timepoints throughout the intervention using SenseWear armband activity monitors and/or Personal Activity IntelligenceTM (using heart rate monitors and smart phone application).
Health-Related Quality of Life | 7 weeks
  Using the Short-Form 36 survey and Satisfaction with Physical Function and Appearance Survey

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No